CLINICAL TRIAL: NCT03853668
Title: Sleep Quality Response to Resisted Training After Coronary Artery Bypass Grafting
Acronym: exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hady Atef Labib, Assistant lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sleep and exercise
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Sleep Deprivation
Keywords: sleep quality; aerobic and resisted exercises; CABG
MeSH Terms: conditions — Sleep Deprivation; Sleep Initiation and Maintenance Disorders | interventions — Exercise; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise group (Active Comparator): aerobic exercises (intervention) on treadmill for 10 weeks, 3 times/week for duration of 30-45 min/session.
  Exercise intensity is 50-65%of maximal heart rate (MHR)
  Interventions: Behavioral: exercise
- aerobic and resisted exercise (Experimental): combined resisted and aerobic exercises (intervention) for 10 weeks (circuit weight training and treadmill training respectively) 2 times/week for a duration of 30-45 min/session Exercise intensity is 50-65%of maximal heart rate (MHR) for aerobic part and 50% of 1 repetition maximum (1RM) for resistance part.
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — control group (n=40) did aerobic exercises on treadmill for 10 weeks experimental group (n=40) did combined aerobic and resisted exercises for 10 weeks
  Other Names: cardiac rehabilitation

SUMMARY:
Background:There are still many gaps in research concerning the effect of different physical training modalities on sleep quality in the population underwent coronary artery bypass graft surgeries(CABG).Purpose:The present study was conducted to compare the quality of sleep in subjects who underwent CABG, were submitted to two types of training (i.e, aerobic exercise alone or combined aerobic and resistance training

DETAILED DESCRIPTION:
OBJECTIVE/BACKGROUND:

There are still many gaps in research concerning the effect of different physical training modalities on sleep quality in the cardiac population. Thus, the objective of the present study was to compare the quality of sleep in subjects who underwent coronary artery bypass surgery submitted to two types of training (ie, aerobic exercise alone or combined aerobic and resistance training).

PATIENTS/METHODS:

80 Participants aged 45-65 years were randomized to two groups: aerobic group (AG), combined aerobic and resistance group (ARG). Training lasted ten consecutive weeks with 30 uninterrupted sessions. The actigraph (Actiwatch Minimitter Company, Incorporated (INC) - Sunriver, OR, USA) was placed on the non-dominant wrist and activities were monitored continuously while being recorded at one minute intervals. The participants kept the device for a period of 96 hours before the first and last training sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have underwent CABG surgery since 6-8 weeks
2. Their ages ranges from 40 and 80 years of age
3. Medically stable patients.
4. patients did CABG-only treatment (not combined with valve replacement surgery)
5. Current complaint of poor Sleep quality (SQ) (score > 5 of the SQ scale)
6. Body mass index ≤ 35 kg/m2 (no obstructive sleep apnea)

Exclusion Criteria:

1. Any patient is known to have any unstable medical condition
2. History of chronic insomnia for at least one year before surgery
3. Indication of receiving treatments for depression and anxiety
4. Musculoskeletal or neurological conditions that might interfere with the execution or the assessment of the exercise.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
sleep quality to be assessed by Pittsburgh Sleep Quality Index (PSQI) | up to 12 months
  1.The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval.
sleep fragmentation index to be assessed by actigraphy | up to 12 months
  2.Actigraphy is a valid tool to assist in determining sleep patterns in normal, healthy adult populations, normal infants and children, and patients suspected of certain sleep disorders.

SECONDARY OUTCOMES:
Functional aerobic capacity to be assessed by 6 minute walk test (6MWT) | 6 months
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Hady Atef, Master, Principal Investigator — Assistant lecturer of physical therapy,Cairo University
Locations (1):
- National heart institute, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided